CLINICAL TRIAL: NCT02244112
Title: A Phase 1 Study of Oprozomib to Assess Food Effect, Drug-Drug Interaction With Midazolam, and Safety and Tolerability in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Why study stopped revised to "A program evaluation identified that the safety profile and pharmacokinetic (PK) characteristics of the formulation used in all oprozomib studies required further optimization and thus enrollment in OPZ009 was halted
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPZ009
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2018-04

CONDITIONS: Advanced Non-Central Nervous System (CNS) Malignancies
MeSH Terms: conditions — Neoplasms | interventions — ONX 0912; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part I: Food Effect/QTc (Experimental): Subjects will receive a single dose of oprozomib 270 mg in 1 of 3 fasting/fed conditions:
  * Diet A: Fasted conditions
  * Diet B: A low-fat breakfast. A low-fat breakfast is defined as having a total caloric value of less than 400 calories, with less than 20% from fat
  * Diet C: A high-fat breakfast. A high-fat breakfast is defined as having a total caloric value of 800 to 1000 calories, with approximately 50% from fat
  Interventions: Drug: Oprozomib
- Part II: Drug-Drug Interaction (DDI) (Experimental): * Period 1: Midazolam 2 mg single oral dose on one day between Day -7 and -4
  * Period 2: Midazolam 2 mg single oral dose 1 hour following oprozomib dose on Day 1 of Cycle 1 and Day 2 of Cycle 2. Oprozomib 300 mg dose on Days 1, 2, 8 and 9 of Cycles 1 and Cycle 2
  Interventions: Drug: Oprozomib; Drug: Midazolam
- Extension (Experimental): After subjects complete the Food Effect/QTc or DDI part, subjects may participate in the extension part of the study, where oprozomib treatment will be continued on Days 1, 2, 8, and 9 of each 14-day cycle. During this part of the study, it is recommended that oprozomib be taken with food.
  Interventions: Drug: Oprozomib

INTERVENTIONS:
Drug: Oprozomib — Subjects will receive oprozomib 270 mg per dose in Part I and oprozomib 300 mg per dose in Part II.
Drug: Midazolam — Subjects will receive a single oral dose of midazolam 2 mg in Period 1 and oral midazolam 2 mg per dose in Period 2.
  Arms: Part II: Drug-Drug Interaction (DDI)

SUMMARY:
The purpose of this Phase 1 of the study is to evaluate the effect of food on the pharmacokinetics (PK) of oprozomib, the drug-drug interaction of oprozomib with midazolam, and the safety and tolerability of oprozomib in patients with advanced malignancies

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of an advanced malignancy.
2. Relapsed after standard therapy for their malignancy, or if no standard therapy is defined, relapsed after investigational therapy and considered by the treating physician to be an appropriate candidate for a Phase 1 clinical study
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
4. Adequate hepatic function, with bilirubin ≤ 1.5 times the upper limit of normal (ULN) in the absence of Gilbert's disease or hemolysis, and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times ULN.
5. Absolute neutrophil count (ANC) ≥ 1000/mm3. Screening ANC must be independent of myeloid growth factor support for at least 1 week, or pegylated growth factors for 2 weeks.
6. Hemoglobin > 7g/dL. Patients may receive red blood cell (RBC) transfusions or erythropoietin or darbepoetin in accordance with institutional guidelines up to 1 week before screening.
7. Platelet count > 30,000 mm3. Patients will not have received platelet transfusions for at least 1 week before screening.
8. Uric acid, if elevated, must be lowered to less than the ULN.
9. Calculated or measured creatinine clearance (CrCl) ≥ 30 mL/min calculated using the formula of Cockcroft and Gault [(140 - age) × mass (kg) / (72 × serum creatinine mg/dL)]. Multiply result by 0.85 if female.

Key Exclusion Criteria:

1. Recovered (i.e., ≤ Grade 1 toxicity or patient's baseline status) from the reversible nonhematologic effects of prior anticancer therapy, excluding alopecia.
2. Systemic chemotherapy with approved or investigational anticancer therapeutics, including steroid therapy intended to treat underlying malignancy, within 3 weeks before the first oprozomib dose; for antibody therapy, a minimum of 3 half-lives must elapse before the first oprozomib dose.
3. Radiation therapy within 3 weeks before first oprozomib dose. Radioimmunotherapy within 8 weeks before first oprozomib dose.
4. Autologous stem cell transplant (ASCT) within 8 weeks and allogeneic SCT within 16 weeks prior to initiation of study treatment. Patients with prior allogeneic SCT must not have evidence of moderate-to-severe graft-versus-host disease (as defined in Filipovich 2005).
5. Unresolved toxicity (NCI-CTCAE version 4.03) ≥ Grade 2 from previous anticancer therapy, except alopecia.
6. Major surgery within 3 weeks before first oprozomib dose.
7. Congestive heart failure (New York Heart Association Class III to IV)
8. Symptomatic cardiac ischemia.
9. Conduction abnormalities uncontrolled by conventional intervention, including but not limited to persistent or permanent atrial fibrillation.
10. History of ventricular fibrillation or ventricular tachycardia.
11. History of torsade de pointe.
12. Myocardial infarction within 6 months before first dose.
13. Abnormal measurements on 12-lead ECG.
14. Uncontrolled diabetes mellitus or hypertension
15. Dysphagia or inability to swallow tablets.
16. Insufficiency of the exocrine pancreas, steatorrhea, or other disorders of the digestive system that impair absorption.
17. Resection of any portion of the stomach or intestines, with the exception of appendectomy.
18. History of bariatric surgery, except in cases where no bowel was resected and all devices have been removed.
19. Active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks before first dose, unless cultures or polymerase chain reaction (PCR) have been negative for 14 days.
20. Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive, or suspected hepatitis C infection.
21. Primary malignancy of the central nervous system.
22. Patient has symptomatic brain metastasis. Patients with brain metastases must have stable neurologic status following surgery or radiation for at least 2 weeks after completion of the definitive therapy, AND be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
23. Significant peripheral neuropathy (Grade 2 with pain or ≥ Grade 3).
24. Systemic treatment with strong inhibitors of P-glycoprotein ([P-gp]; i.e., itraconazole, ketoconazole) within 14 days before the first dose of oprozomib.
25. Patients must not have used any potent CYP3A4 inhibitors (i.e., ketoconazole) within 7 days prior to enrollment, or any potent CYP3A4 inducers (i.e., rifampin) within 14 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05-15 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Food Effect/QTc - Cmax | Approximately 5 days or up to 2 weeks
  Pharmacokinetics (PK) parameter Cmax (maximum plasma concentration of oprozomib) between each diet (oprozomib under fasting versus low-fat, and fasting versus high-fat conditions).
Food Effect/QTc - AUC | Approximately 5 days or up to 2 weeks
  Pharmacokinetics (PK) parameter AUC (area under the concentration-time curve from time zero to the last measurable time point [AUC0-t], area under the concentration-time curve from time zero to infinity [AUC0-inf]) of oprozomib between each diet (oprozomib under fasting versus low-fat, and fasting versus high-fat conditions).
Food Effect - tmax and t1/2 | Approximately 5 days or up to 2 weeks
  Pharmacokinetics (PK) parameters tmax (time to reach maximum plasma concentration) and t1/2 (terminal half-life) between each diet (oprozomib under fasting versus low-fat, and fasting versus high-fat conditions).
Food Effect - QT/QTc interval | Approximately 5 days or up to 2 weeks
  QT/QTc interval will be extracted from continuous ECGs performed during each period in the Food Effect/QTc part of the study:
  * Twelve (12)-lead ECGs will be serially recorded digitally and read centrally
  * The RR, PR and QT intervals and QRS duration will be analyzed
  * QTc will be calculated using Bazett's and Fridericia's formulas
Drug-Drug Interaction (DDI) - Cmax | Approximately 1 month
  Pharmacokinetics (PK) parameter Cmax (maximum plasma concentration) of midazolam, in the presence and absence of oprozomib.
Drug-Drug Interaction (DDI) - AUC | Approximately 1 month
  Pharmacokinetics (PK) parameter AUC (area under the concentration-time curve from time zero to the last measurable time point [AUC0-t], area under the concentration-time curve from time zero to infinity [AUC0-inf]) of midazolam, in the presence and absence of oprozomib.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 18 months
  Number of patients that experience Adverse Events (AEs). Adverse Events (AEs) and Serious Adverse Events (SAEs) graded according to the NCI-CTCAE (Version 4.03).

OTHER OUTCOMES:
Overall Response Rate (ORR) | Approximately 18 months
  Overall Response Rate (ORR) according to disease-specific response criteria
Time To Progression (TTP) | Approximately 18 months
  Time to progression (TTP) according to disease-specific evaluation criteria

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Winship Cancer Institute, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Mary Crowley Cancer Research Centers - Medical City, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah